CLINICAL TRIAL: NCT01495949
Title: The Changes in Cortisol Levels and Stress Responses During Cardiac Surgery. The Comparison Between Two Induction Agents: Etomidate and Thiopentone.
Brief Title: The Cortisol Levels During Cardiac Surgery. The Comparison Between Etomidate and Thiopentone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Manee Raksakietisak, Associate professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si559/2011
Record Dates: First submitted 2011-12-13; First posted 2011-12-20 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease
Keywords: etomidate; cortisol level; inotrope; cardiac patients
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases | interventions — Etomidate; Thiopental

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- etomidate (Active Comparator)
  Interventions: Drug: etomidate
- thiopentone (Active Comparator)
  Interventions: Drug: thiopentone

INTERVENTIONS:
Drug: etomidate — During induction, after 3 mcg/kg of fentanyl and 0.05 mg/kg of midazolam given, small doses 2-4 mg (1-2 ml) of etomidate will be given by titration (the syringe pump and extension and three way stopcock are covered to blind the study drug) until the patients are unconscious.
  Other Names: Etomidate Lipuro (B Braun company)
  Arms: etomidate
Drug: thiopentone — During induction, after 3 mcg/kg of fentanyl and 0.05 mg/kg of midazolam given, small doses 25-50 mg (1-2 ml) of thiopentone will be given by titration (the syringe pump and extension and three way stopcock are covered to blind the study drug) until the patients are unconscious
  Other Names: Anesthal (Jagsonpal pharmaceuticals Ltd)
  Arms: thiopentone

SUMMARY:
During induction for cardiac surgery, patient hemodynamic stability is achieved by using anesthetic drugs which least affects hemodynamics such as benzodiazepines, etomidate. Etomidate although has been used for a long time but its safety regarding cortisol synthesis suppression is still doubtful. This study measures the changes in cortisol levels during cardiac surgery with the use of cardiopulmonary bypass by comparison between two inductive agents (etomidate and thiopentone). Recording data also include hemodynamic changes during induction, inotropic use for coming of cardiopulmonary bypass, blood glucose levels, amount of insulin usage, length of ICU and hospital saty.

DETAILED DESCRIPTION:
Ninety-two cardiac patients who undergoing cardiopulmonary bypass graft (CABG) or valve surgery will be enrolled in this study. They will be randomized into two groups (thiopentone and etomidate groups). Apart from different in two inductive drugs, other anesthetics will be the same. We record hemodynamic changes during inductions, inotropic use (dose and duration), blood glucose levels, total insulin requirement to keep blood glucose 140-180 mg% in perioperative period, duration of mechanical ventilation, length of stay in ICU and total hospital length of stay. The changes in cortisol levels will be recorded at time 0 (before induction), 2, 4, 8, 24 hours in 26 patients (13 patients in each group and only patients who are the first in the operating list (morning list)).The 26 patients is needed from sample size equation for the changes in cortisol level and the 92 patients is calculated from the differences in inotropic use.

ELIGIBILITY:
Inclusion Criteria:

60 year or older cardiac patient undergoing cardiac surgery (CABG or valve surgery) with the use of cardiopulmonary bypass -

Exclusion Criteria:

* Redo or emergency operation
* complex and prolong operation
* history of adrenal insufficiency or steroid use
* already has inotropic drugs to support hemodynamics
* creatinine > 2.0 mg/dl

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
cortisol levels | baseline (before induction), 2, 4, 8, and 24 hrs
  Measure cortisol levels and its changes due to stress response during surgery. Compare the changes in cortisol levels between two induction agents (etomidate and thiopentone).

SECONDARY OUTCOMES:
the use of inotropes for maintaining hemodynamic | 24 hours
  The dose and duration of inotropic drug (S) used for maintaining hemodynamic during coming off cardiopulmonary bypass and postoperative period.
Length of ICU and hospital stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Manee Raksakietisak, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital Mahidol University, Bangkok, Thailand

REFERENCES:
- [Derived] Raksakietisak M, Ngamlamiad C, Duangrat T, Soontarinka S, Raksamani K. The Changes in Cortisol Levels during Cardiac Surgery: A Randomized Double-Blinded Study between Two Induction Agents Etomidate and Thiopentone. J Med Assoc Thai. 2015 Aug;98(8):775-81. PMID 26437535